CLINICAL TRIAL: NCT03335904
Title: Effect of Angiotensin Receptor Blockers on Periodic Breathing During Sleep in Hypoxia
Brief Title: AT1R Blockade and Periodic Breathing During Sleep in Hypoxia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Glen Foster, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H17-02920
Record Dates: First submitted 2017-11-01; First posted 2017-11-08 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Sleep Disordered Breathing; Hypoxia; Respiration; Sleep Disorder; Chemoreceptor Apnea
Keywords: Angiotensin receptor blockade; control of breathing; breath-holding
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypoxia; Respiratory Aspiration; Sleep Wake Disorders | interventions — Losartan; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will ingest microcrystalline cellulose by mouth on two consecutive days. The first tablet will be consumed on day 1 at 0700 hrs. The second tablet will be consumed at 1900 hrs and the final tablet will be consumed at 0700hrs on day 2. Participants will undergo a Hyperoxic Hypercapnic Ventilatory Response Test, a Hypoxic Hypercapnic Ventilatory Response Test, and Repeated Hypoxic Apneas before and after a Hypoxic Sleep Study.
  Interventions: Other: Hyperoxic Hypercapnic Ventilatory Response Test; Other: Hypoxic Hypercapnic Ventilatory Response Test; Other: Repeated Hypoxic Apneas; Other: Hypoxic Sleep Study; Drug: Placebo
- Losartan (Experimental): Participants will ingest 50 mg of losartan, an angiotensin receptor blocker, by mouth on two consecutive days. The first tablet will be consumed on day 1 at 0700 hrs. The second tablet will be consumed at 1900 hrs and the final tablet will be consumed at 0700hrs on day 2. Participants will undergo a Hyperoxic Hypercapnic Ventilatory Response Test, a Hypoxic Hypercapnic Ventilatory Response Test, and Repeated Hypoxic Apneas before and after a Hypoxic Sleep Study.
  Interventions: Other: Hyperoxic Hypercapnic Ventilatory Response Test; Other: Hypoxic Hypercapnic Ventilatory Response Test; Other: Repeated Hypoxic Apneas; Other: Hypoxic Sleep Study; Drug: Losartan

INTERVENTIONS:
Other: Hyperoxic Hypercapnic Ventilatory Response Test — End-tidal PO2 will be clamped at 300 mmHg while end-tidal PCO2 will be increased in three minutes stages from baseline to +2, +4, and +6 mmHg.
Other: Hypoxic Hypercapnic Ventilatory Response Test — End-tidal PO2 will be clamped at normoxic levels while end-tidal PCO2 will be increased in three minutes stages from baseline to +2, +4, and +6 mmHg.
Other: Repeated Hypoxic Apneas — Six hypoxic apnea cycles will be performed. One apneic cycle involves breathing 2-3 breaths of 100% Nitrogen and breath-holding for 20s followed by room air breathing.
Other: Hypoxic Sleep Study — Participants will be instrumented with a sleep monitoring system and will sleep in a normobaric hypoxic chamber with a fraction of inspired oxygen of 13.5%.
Drug: Losartan — Losartan, 50mg, BID
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — Placebo, 50mg, BID
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
Sleep disordered breathing (SDB) is characterized by regular periods of no breathing (apnea) or low levels of breathing (hypopnea) and leads to repeated periods of low oxygenation, termed intermittent hypoxia that causes fluctuations in blood oxygen levels. This leads to increased peripheral chemoreflex sensitivity that is thought to occur through the stimulation of angiotensin-II, type-I receptors (AT1R) that are expressed primarily on glomus cells within the peripheral chemoreflex and ultimately results in long lasting hypertension. The goal of this study is to determine if AT1R receptor blockade can prevent the increase in chemoreflex sensitivity following one night of hypoxia and improve the severity of SDB.

DETAILED DESCRIPTION:
Objective: To determine the effects of angiotensin-II, type-I receptor (AT1R) blockade on the relationship between ventilatory control and sleep disordered breathing (SDB) following a night of hypoxic sleep in healthy humans.

Justification: Ventilatory adaptation to hypoxia is one of two major adaptations permitting humans to acclimatize successfully to high altitude. As the partial pressure of oxygen falls with ascent, the peripheral chemoreceptors are stimulated resulting in an increase in ventilation. The initial hypoxic ventilatory response is aimed at augmenting alveolar PO2 and subsequently arterial PO2, but results in a respiratory alkalosis that can only be compensated for by the reduction of renal excretion of bicarbonate. Despite metabolic compensation, both basal respiratory drive and peripheral chemoreceptor responsiveness remain elevated. Both of these elements of respiratory control have contrasting implications for breathing stability during sleep. The increase in basal ventilation at high altitude attenuates plant gain, a term describing how effectively a change in ventilation changes blood gases. Plant gain is determined by positioning the chemoreflex response on the isometabolic hyperbola. When arterial PCO2 is reduced during acclimatization to high altitude, the point of equilibrium is shifted to a steeper portion of the isometabolic hyperbola where a larger change in ventilation is necessary to evoke a given change in arterial PCO2. This feature is protective in nature and acts to stabilize breathing. However, the slope of the relationship between ventilation and arterial PCO2, termed controller gain, is greatly enhanced at high altitude and this may outweigh the effect on plant gain, destabilizing breathing and predisposing to central sleep apnea. Treatments that reduce controller gain without impacting plant gain might stabilize breathing and reduce the severity of central sleep apnea at high altitude without negatively impacting successful acclimatization.

The carotid body chemoreceptors serve an important regulatory role in controlling alveolar ventilation and their sensitivity is augmented at high altitude. Recent studies have established that the carotid body possesses a local angiotensin system, which contributes to the sensitization of the chemoreflex function in patients with heart failure, sleep apnea, and following exposure to intermittent hypoxia. Indeed, the over-activity of the carotid body contributes to breathing instability and increases the incidence of central apneas. Angiotensin II activates the carotid body and leads to afferent activity. The Type I cells within the carotid body act as a chemical sensor and they express both angiotensinogen and express two angiotensin receptors, AT1R and AT2R. Interestingly, pharmacological blockade of the AT1R has little functional significance at sea level in the normal state. But if chemoreceptor activity is augmented in conditions such as chronic, and intermittent hypoxia, and congestive heart failure, then blockade of the AT1R partially reverses this activity. Whether or not AT1R blockade at high altitude can attenuate the rise in chemoreceptor sensitivity and reduce the severity of sleep apnea in humans is unknown.

Purpose: To determine if blockade of the AT1R can attenuate the ventilatory response to CO2 and reduce the severity of sleep disordered breathing in healthy humans.

Hypothesis: Blockade of the AT1R will reduce the ventilatory sensitivity to CO2 and the severity of SDB in healthy humans following one night of hypoxia.

Research Design General Procedures: Sleep studies will be conducted between 2100hrs and 0600 hrs. Participants will arrive at the laboratory in the evening and will be allowed to sleep in the hypoxic chamber for 8 hours. Ventilatory responses will be assessed prior to entering the hypoxic chamber and immediately upon waking in the morning following sleep study. Either Losartan, an AT1R antagonist, (50 mg/dose; P.O.) or placebo will be administered three times throughout the protocol: the morning of the experimental day, the evening one hour prior to the ventilatory tests and finally the following morning after a night in the hypoxic chamber, one hour prior to the second battery of ventilatory tests. This protocol design is randomized, double blinded and placebo controlled and all participants will complete both experimental arms separated by at least 2 days (i.e. cross-over study design). During the ventilatory tests, participants will be studied in the supine position, 6 hours post-prandial & 24 hours post-caffeine, and breathing through a standard mouthpiece with a nose clamp. Non-invasive measures of heart rate (HR), blood pressure (BP), respiratory frequency (fB), tidal volume (VT), minute ventilation (V̇E), cerebral blood flow [assessed by transcranial Doppler (MCA and PCA)], end-tidal gases (PETCO2 and PETO2) and blood oxygen saturation (SpO2; finger pulse oximetry) will be monitored and recorded continuously. Venipuncture will be performed immediately prior to both ventilatory response tests and will be analyzed for plasma renin activity levels to confirm functional angiotensin receptor blockade.

ELIGIBILITY:
Inclusion Criteria:

* normotensive
* forced expiratory volume in 1s : forced vital capacity ratio > 0.75
* no medical history of cardiovascular and respiratory disease
* not taking medications other than oral contraceptives
* free from sleep apnea
* body mass index less than 30 kg/m2

Exclusion Criteria:

* history of hypertension
* known impaired renal function
* liver disease
* heart failure
* myocardial infarction
* coronary artery disease
* smoked within the past year
* apnea hypopnea index > 5 events per hour

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
apnea-hypopnea index | 8 hours
  the number of apnea and hypopneas per hour during sleep in hypoxia

SECONDARY OUTCOMES:
Average oxygen saturation | 8 hours
  average oxyhemoglobin saturation measured during sleep in hypoxia
Hyperoxic Hypercapnic Ventilatory Response | 0 and 8 hours
  The change in ventilation per change in end-tidal PCO2 measured in a background of hyperoxia
Hypoxic Hypercapnic Ventilatory Response | 0 and 8 hours
  The change in ventilation per change in end-tidal PCO2 measured in a background of hypoxia
Change in systolic and diastolic blood pressure during breath-hold | 0 and 8 hours
  The blood pressure response to repeated 20s hypoxic breath-holds.
Hyperoxic Hypercapnic Cerebral Blood Flow Response | 0 and 8 hours
  the change in middle cerebral and posterior cerebral blood velocity per change in end-tidal PCO2 measured in a background of hyperoxia
Hypoxic Hypercapnic Cerebral Blood Flow Response | 0 and 8 hours
  the change in middle cerebral and posterior cerebral blood velocity per change in end-tidal PCO2 measured in a background of hypoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Glen Foster, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

REFERENCES:
- [Result] Brown CV, Boulet LM, Vermeulen TD, Sands SA, Wilson RJA, Ayas NT, Floras JS, Foster GE. Angiotensin II-Type I Receptor Antagonism Does Not Influence the Chemoreceptor Reflex or Hypoxia-Induced Central Sleep Apnea in Men. Front Neurosci. 2020 Apr 28;14:382. doi: 10.3389/fnins.2020.00382. eCollection 2020. PMID 32410951